CLINICAL TRIAL: NCT04154579
Title: A Randomized Controlled Trial Utilizing the Arts to Improve Health, Resilience, and Well-Being in Individuals With Chronic Health Conditions in Underserved Neighborhoods
Brief Title: Arts & Health Education to Improve Health, Resilience, and Well-Being
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic. Unable to restart as had hoped.
Sponsor: Lisa Gallagher (Other)
Collaborators: National Endowment for the Arts, United States (U.S. Federal Agency); Cuyahoga Arts and Culture (Unknown); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Lisa Gallagher, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#19-854
Record Dates: First submitted 2019-10-02; First posted 2019-11-06 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Hypertension; Diabetes; Obesity; COPD; CHF; High Cholesterol; Asthma; Chronic Pain; Multiple Sclerosis; Depression; Anxiety; Heart Diseases; Stroke
Keywords: Chronic health conditions; Arts-based program; Health education program; Health; Resilience; Well-being
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Obesity; Pulmonary Disease, Chronic Obstructive; Hypercholesterolemia; Asthma; Chronic Pain; Multiple Sclerosis; Depression; Anxiety Disorders; Heart Diseases; Stroke | interventions — Music Therapy; Art Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial utilizing a mixed methods, pre-post intervention, and parallel group analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HeRe We Arts (Experimental): This is an 8 week, arts-based session that includes educational & experiential components. Topics include: Introduction to Arts & Health; Music, Well-Being, & Resilience; Movement & Physical Activity; Art & Well-Being; Writing & Communication/Self-Expression; Theater & Socialization; Art Appreciation & a Healthy Brain; & Summary/Integration of the Arts into Daily Lives.
  Interventions: Behavioral: HeRe We Arts
- HeRe We Ed (Health Education Group) (Active Comparator): This is an 8 week, non-arts-based health education session that includes educational & some experiential components. Topics include: Introduction to Health, Resilience, & Well-Being; Nutrition & Healthy Eating; Exercise, Chair Yoga, & Sleep; Mental Health, Stress Management, & Life Satisfaction; Holistic Approaches: Wellness, Integrative Medicine, & Complementary & Alternative Medicine; Chronic Illnesses & Chronic Pain; Health & Behaviors; Summary & Navigating the Healthcare System.
  Interventions: Behavioral: HeRe We Ed

INTERVENTIONS:
Behavioral: HeRe We Arts — Art Therapy interventions to promote health, resilience & well-being will discussed; & experiences such as key chain making, collaging on journal covers, creating sculpture garden will be utilized. Music therapy interventions such as lyric discussion, singing, instrument playing, & music-assisted relaxation techniques will be utilized; & discussion of use of music to elicit positive physical & emotional responses will be held. Drums Alive (drumming & movement) will be used to promote physical activity. Art appreciation will include discussion of public art forms. Journaling will include different techniques for journaling, writing poetry, etc. Theater games such as Password, Press Conference, Props Only, & Draw What You Hear will be utilized. Chair yoga will be introduced as a form of exercise. Education will be provided on the various topics.
  Other Names: Music Therapy; Drums Alive; Art Appreciation; Journaling; Theater Games; Art Therapy
  Arms: HeRe We Arts
Behavioral: HeRe We Ed — Educational components and some experiential components will be utilized to educate the participants on health, resilience, well-being, nutrition, healthy eating, weight management, eating disorders, obesity, exercise, physical activity, sleep hygiene and the importance of sleep, mental health, stress management, the importance of improving life satisfaction, holistic approaches, wellness, integrative medicine, complementary and alternative medicine, chronic illness, chronic pain, methods for dealing with chronic versus acute illnesses, changing behaviors and/or maintaining healthy behaviors in order to promote health and stay out of the hospital, and navigating the healthcare system. Specific experiential components will include Chair Yoga and Stress Management Techniques.
  Other Names: Health Education; Chair Yoga; Stress Management Techniques
  Arms: HeRe We Ed (Health Education Group)

SUMMARY:
This is an 8-week randomized controlled trial to help address health, resilience, and well-being. Participants are randomized into either a health education group or an arts-based health education group. Both groups will attend for 8 weeks and various study assessments will be conducted in order to measure the experience and impact of the program. Anyone 18 years and older with a chronic health condition (for example, diabetes, hypertension, congestive heart failure, chronic obstructive pulmonary disorder, asthma, weight, anxiety, depression, cardiac, arthritis, multiple sclerosis, and many more) are eligible to participate.

DETAILED DESCRIPTION:
Within the healthcare field today there is an increased concern with public health, population health, wellness, and prevention, all of which include focusing on physical health, obesity, chronic health conditions, unhealthy lifestyles, aging, and mental health issues. As healthcare professionals attempt to improve individuals' health outcomes, quality of life, well-being, coping skills, and health indicators, they also must try to promote behavior change that helps keep patients out of the hospital. These are concerns faced by individuals of all ages, genders, ethnicities, cultural backgrounds, socioeconomic statuses, and diagnoses. Therefore, it is important to find multiple means of addressing these concerns with the various populations as it is likely that no one particular method would be effective for every individual.

Programs and interventions have been created to address health, resilience, and well-being at the individual and the social level. They demonstrate the importance of providing support, encouraging behavior changes, and reinforcing objectives determined by the healthcare system. Many of these programs have focused on improving resilience and increasing participants' ability to thrive or recover from the illnesses and challenges they face.

The broad problem to be addressed by this study is to assess if arts-based programs are superior to non-arts-based health education programs at improving individuals' physical and mental health outcomes, quality of life, well-being, resilience, coping skills, stress, and health indicators while promoting behavior change and keeping them out of the hospital. Previous programs have focused on improving resilience. Individual arts interventions such as music, art, craft, choir singing, writing, theater, and movement have been utilized and in many cases found to be helpful in addressing resilience, coping, health, and well-being; however, it is not known what effect a program utilizing multiple arts-based interventions would have on adults with chronic health conditions. The primary benefit of conducting research into the effectiveness of different arts-based programs is the identification of the specific benefits of programs aimed at influencing health, resilience, and well-being in individuals with a variety of chronic health conditions.

The purpose of this randomized controlled study is to determine the outcomes of an 8-week arts-based program on the health, resilience, and well-being of individuals with chronic health conditions in an outpatient underserved community setting as compared to outcomes from individuals participating in a separate 8-week-non-arts-based health education program in the same setting. The purpose of including a variety of arts experiences is so that individuals will hopefully find at least one art form to which they can relate and will utilize in their lives to assist with their health, resilience, and well-being. The non-arts-based program will include educational topics related to health, resilience, and well-being.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnosed with at least one chronic health condition (as reported by the participant)
* Able to participate safely in all program sessions
* Proficient in English
* Cognitively able to consent to participate

Exclusion Criteria:

* Severe visual or auditory impairment
* Severe and/or uncontrolled comorbidity precluding safe participation in the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Change in Short Depression-Happiness Scale from Week 1 to Week 8 | Weeks 1 and 8
  Means of assessing change in mood. Contains 6 items, 3 negative & 3 positive. Participants think about how they felt in the past 7 days & rate the frequency of each item on a 4-point scale. Scale ranges include scores between 0 and 18. Higher scores indicate higher levels of happiness.
Change in Short Depression-Happiness Scale from Week 8 to Week 16 | Weeks 8 and 16
  Means of assessing change in mood. Contains 6 items, 3 negative & 3 positive. Participants think about how they felt in the past 7 days & rate the frequency of each item on a 4-point scale. Scale ranges include scores between 0 and 18. Higher scores indicate higher levels of happiness.
Change in Short Depression-Happiness Scale from Week 1 to Week 16 | Weeks 1 and 16
  Means of assessing change in mood. Contains 6 items, 3 negative & 3 positive. Participants think about how they felt in the past 7 days & rate the frequency of each item on a 4-point scale. Scale ranges include scores between 0 and 18. Higher scores indicate higher levels of happiness.
Change in Short Warwick-Edinburgh Mental Well-Being Scale from Week 1 to Week 8 | Weeks 1 and 8
  Participants answer 7 questions by choosing the answer that best describes their experience over the last 2 weeks. Designed to measure the feeling and functioning aspects of positive mental well-being. Scores range from 7 to 35. Higher scores represent higher positive mental well-being.
Change in Short Warwick-Edinburgh Mental Well-Being Scale from Week 8 to Week 16 | Weeks 8 and 16
  Participants answer 7 questions by choosing the answer that best describes their experience over the last 2 weeks. Designed to measure the feeling and functioning aspects of positive mental well-being. Scores range from 7 to 35. Higher scores represent higher positive mental well-being.
Change in Short Warwick-Edinburgh Mental Well-Being Scale from Week 1 to Week 16 | Weeks 1 and 16
  Participants answer 7 questions by choosing the answer that best describes their experience over the last 2 weeks. Designed to measure the feeling and functioning aspects of positive mental well-being. Scores range from 7 to 35. Higher scores represent higher positive mental well-being.
Change in Brief Resilient Coping Scale from Week 1 to Week 8 | Weeks 1 and 8
  A 4-item measure designed to identify participants' abilities to cope with stress. It may be helpful for recognizing those who may need to learn techniques to help improve their coping skills and resilience. Scores range from 4-20. Scores of 4-13 represent low resilient copers, those of 14-16 represent medium resilient copers, and those of 17-20 represent high resilient copers.
Change in Brief Resilient Coping Scale from Week 8 to Week 16 | Weeks 8 and 16
  A 4-item measure designed to identify participants' abilities to cope with stress. It may be helpful for recognizing those who may need to learn techniques to help improve their coping skills & resilience. Scores range from 4-20. Scores of 4-13 represent low resilient copers, those of 14-16 represent medium resilient copers, and those of 17-20 represent high resilient copers.
Change in Brief Resilient Coping Scale from Week 1 to Week 16 | Weeks 1 and 16
  A 4-item measure designed to identify participants' abilities to cope with stress. It may be helpful for recognizing those who may need to learn techniques to help improve their coping skills & resilience. Scores range from 4-20. Scores of 4-13 represent low resilient copers, those of 14-16 represent medium resilient copers, and those of 17-20 represent high resilient copers.
Change in Godin-Shephard Leisure-Time Physical Activity Questionnaire from Week 1 to Week 8 | Weeks 1 and 8
  Measures amount of physical activity. Asks participants how many times on average, over a 7-day period, they engage in strenuous, moderate, or mild exercise for more than 15 minutes, and the average frequency of activity that leads to increased heart rate. Scores range from 0-24. Higher scores indicate higher levels of physical activity.
Change in Godin-Shephard Leisure-Time Physical Activity Questionnaire from Week 8 to Week 16 | Weeks 8 and 16
  Measures amount of physical activity. Asks participants how many times on average, over a 7-day period, they engage in strenuous, moderate, or mild exercise for more than 15 minutes, and the average frequency of activity that leads to increased heart rate. Scores range from 0-24. Higher scores indicate higher levels of physical activity.
Change in Godin-Shephard Leisure-Time Physical Activity Questionnaire from Week 1 to Week 16 | Weeks 1 and 16
  Measures amount of physical activity. Asks participants how many times on average, over a 7-day period, they engage in strenuous, moderate, or mild exercise for more than 15 minutes, and the average frequency of activity that leads to increased heart rate. Scores range from 0-24. Higher scores indicate higher levels of physical activity.
Change in PROMIS Scale v1.2 - Global Health from Week 1 to Week 8 | Weeks 1 and 8
  A self-report measure to identify symptoms, feelings, behaviors, & functions in the areas of physical, mental, & social health. Raw scores for mental health and for physical health are translated into T-scores. The mean for the T-score is 50 and there is a standard deviation of 10. Therefore, a higher T-score represents higher physical health or higher mental health.
Change in PROMIS Scale v1.2 - Global Health from Week 8 to Week 16 | Weeks 8 and 16
  A self-report measure to identify symptoms, feelings, behaviors, & functions in the areas of physical, mental, & social health. Raw scores for mental health and for physical health are translated into T-scores. The mean for the T-score is 50 and there is a standard deviation of 10. Therefore, a higher T-score represents higher physical health or higher mental health.
Change in PROMIS Scale v1.2 - Global Health from Week 1 to Week 16 | Weeks 1 and 16
  A self-report measure to identify symptoms, feelings, behaviors, & functions in the areas of physical, mental, & social health. Raw scores for mental health and for physical health are translated into T-scores. The mean for the T-score is 50 and there is a standard deviation of 10. Therefore, a higher T-score represents higher physical health or higher mental health.
Change in Systolic and Diastolic Blood Pressure from Week 1 to Week 8 | Weeks 1 and 8
  At the start of each session an investigator will take and document each participants' systolic and diastolic blood pressure.
Change in Systolic and Diastolic Blood Pressure from Week 8 to Week 16 | Weeks 8 and 16
  At the start of each session an investigator will take and document each participants' systolic and diastolic blood pressure.
Change in Systolic and Diastolic Blood Pressure from Week 1 to Week 16 | Weeks 1 and 16
  At the start of each session an investigator will take and document each participants' systolic and diastolic blood pressure.
Change in Heart Rate from Week 1 to Week 8 | Weeks 1 and 8
  At the start of each session an investigator will take and document each participant's heart rate.
Change in Heart Rate from Week 8 to Week 16 | Weeks 8 and 16
  At the start of each session an investigator will take and document each participant's heart rate.
Change in Heart Rate from Week 1 to Week 16 | Weeks 1 and 16
  At the start of each session an investigator will take and document each participant's heart rate.
Change in Pulse Oximetry from Week 1 to Week 8 | Weeks 1 and 8
  At the start of each session an investigator will take and document each participant's pulse oximetry.
Change in Pulse Oximetry from Week 8 to Week 16 | Weeks 8 and 16
  At the start of each session an investigator will take and document each participant's pulse oximetry.
Change in Pulse Oximetry from Week 1 to Week 16 | Weeks 1 and 16
  At the start of each session an investigator will take and document each participant's pulse oximetry.

SECONDARY OUTCOMES:
Change in HeRe We Arts Survey from Week 1 to Week 8 | Weeks 1 and 8
  A pre-test/post-survey utilized to test knowledge on arts and well-being, as well as satisfaction at endpoints. This is not a standardized measure and does not include a scale. It involves changes in knowledge and use of arts techniques, as well as satisfaction with the program via the use of open-ended and multiple choice questions.
Change in HeRe We Ed Survey from Week 1 to Week 8 | Weeks 1 and 8
  A pre-test/post-test utilized to test knowledge on health education & well-being, as well as satisfaction, at endpoints. This is not a standardized measure and does not include a scale. It involves changes in knowledge and use of arts techniques, as well as satisfaction with the program via the use of open-ended and multiple choice questions.
Weekly Post-Session Survey | Weeks 1-8
  Completed by participants at the end of each session in order to obtain information on learning and satisfaction. This is not a standardized measure and does not include a scale. It involves changes in knowledge and use of arts techniques, as well as satisfaction with the program via the use of open-ended and multiple choice questions.

OTHER OUTCOMES:
Weekly Take-Away Goals | Weeks 1-8
  Participants will identify a goal each week, and the next week they will report on whether or not they completed their goal. This does not include a scale. It is merely a Yes or No.
Phone Interview | Week 9
  Phenomenological interviews will be conducted in order to gather qualitative information regarding participants' experience with the program, as well as its impact and meaning in their lives. This does not include a scale. It involves open-ended, qualitative information that is shared.
HeRe We Arts Week 16 Survey | Week 16
  Survey to determine progress, maintenance, and/or follow through at Week 16 (2 months after completion of the program). This does not involve a scale. It seeks to determine if skills are still being used 16 weeks after the start of the program via the use of open-ended and multiple choice questions.
HeRe We Ed Week 16 Survey | Week 16
  Survey to determine progress, maintenance, and/or follow through at Week 16 (2 months after completion of the program). This does not involve a scale. It seeks to determine if skills are still being used 16 weeks after the start of the program via the use of open-ended and multiple choice questions.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Gallagher, MA, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Euclid Hospital, Euclid, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahern NR, Kiehl EM, Sole ML, Byers J. A review of instruments measuring resilience. Issues Compr Pediatr Nurs. 2006 Apr-Jun;29(2):103-25. doi: 10.1080/01460860600677643. PMID 16772239
- [Background] Beesley K, White JH, Alston MK, Sweetapple AL, Pollack M. Art after stroke: the qualitative experience of community dwelling stroke survivors in a group art programme. Disabil Rehabil. 2011;33(23-24):2346-55. doi: 10.3109/09638288.2011.571333. Epub 2011 Apr 18. PMID 21501042
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Davydov DM, Stewart R, Ritchie K, Chaudieu I. Resilience and mental health. Clin Psychol Rev. 2010 Jul;30(5):479-95. doi: 10.1016/j.cpr.2010.03.003. Epub 2010 Mar 25. PMID 20395025
- [Background] Deshields TL, Heiland MF, Kracen AC, Dua P. Resilience in adults with cancer: development of a conceptual model. Psychooncology. 2016 Jan;25(1):11-8. doi: 10.1002/pon.3800. Epub 2015 Mar 18. PMID 25787828
- [Background] Dingle GA, Williams E, Jetten J, Welch J. Choir singing and creative writing enhance emotion regulation in adults with chronic mental health conditions. Br J Clin Psychol. 2017 Nov;56(4):443-457. doi: 10.1111/bjc.12149. Epub 2017 Jul 18. PMID 28722166
- [Background] Fancourt D, Perkins R, Ascenso S, Carvalho LA, Steptoe A, Williamon A. Effects of Group Drumming Interventions on Anxiety, Depression, Social Resilience and Inflammatory Immune Response among Mental Health Service Users. PLoS One. 2016 Mar 14;11(3):e0151136. doi: 10.1371/journal.pone.0151136. eCollection 2016. PMID 26974430
- [Background] Gallagher LM, Lagman R, Bates D, Edsall M, Eden P, Janaitis J, Rybicki L. Perceptions of family members of palliative medicine and hospice patients who experienced music therapy. Support Care Cancer. 2017 Jun;25(6):1769-1778. doi: 10.1007/s00520-017-3578-y. Epub 2017 Jan 19. PMID 28105524
- [Background] Gallagher LM, Lagman R, Rybicki L. Outcomes of Music Therapy Interventions on Symptom Management in Palliative Medicine Patients. Am J Hosp Palliat Care. 2018 Feb;35(2):250-257. doi: 10.1177/1049909117696723. Epub 2017 Mar 9. PMID 28274132
- [Background] Gloria CT, Steinhardt MA. Relationships Among Positive Emotions, Coping, Resilience and Mental Health. Stress Health. 2016 Apr;32(2):145-56. doi: 10.1002/smi.2589. Epub 2014 Jun 24. PMID 24962138
- [Background] Goubert L, Trompetter H. Towards a science and practice of resilience in the face of pain. Eur J Pain. 2017 Sep;21(8):1301-1315. doi: 10.1002/ejp.1062. Epub 2017 Jun 2. PMID 28573783
- [Background] Khan WU, Moss H. Increasing Public Health Awareness of and Capacity for Arts-Based Therapy in Medicine. JAMA Neurol. 2017 Sep 1;74(9):1029-1030. doi: 10.1001/jamaneurol.2017.1639. No abstract available. PMID 28783804
- [Background] Lesiuk T. The Effect of Mindfulness-Based Music Therapy on Attention and Mood in Women Receiving Adjuvant Chemotherapy for Breast Cancer: A Pilot Study. Oncol Nurs Forum. 2015 May;42(3):276-82. doi: 10.1188/15.ONF.276-282. PMID 25901379
- [Background] Orjasaeter KB, Ness O. Acting Out: Enabling Meaningful Participation Among People With Long-Term Mental Health Problems in a Music and Theater Workshop. Qual Health Res. 2017 Sep;27(11):1600-1613. doi: 10.1177/1049732316679954. Epub 2016 Nov 28. PMID 27899473
- [Background] Petriwskyj A, Parker D, O'Dwyer S, Moyle W, Nucifora N. Interventions to build resilience in family caregivers of people living with dementia: a comprehensive systematic review. JBI Database System Rev Implement Rep. 2016 Jun;14(6):238-73. doi: 10.11124/JBISRIR-2016-002555. PMID 27532659
- [Background] Phinney A, Moody EM, Small JA. The Effect of a Community-Engaged Arts Program on Older Adults' Well-being. Can J Aging. 2014 Sep;33(3):336-45. doi: 10.1017/S071498081400018X. Epub 2014 Aug 11. PMID 25110936
- [Background] Robb SL, Burns DS, Stegenga KA, Haut PR, Monahan PO, Meza J, Stump TE, Cherven BO, Docherty SL, Hendricks-Ferguson VL, Kintner EK, Haight AE, Wall DA, Haase JE. Randomized clinical trial of therapeutic music video intervention for resilience outcomes in adolescents/young adults undergoing hematopoietic stem cell transplant: a report from the Children's Oncology Group. Cancer. 2014 Mar 15;120(6):909-17. doi: 10.1002/cncr.28355. Epub 2014 Jan 27. PMID 24469862
- [Background] Stuckey HL, Nobel J. The connection between art, healing, and public health: a review of current literature. Am J Public Health. 2010 Feb;100(2):254-63. doi: 10.2105/AJPH.2008.156497. Epub 2009 Dec 17. PMID 20019311
- [Background] Swarthout M, Bishop MA. Population health management: Review of concepts and definitions. Am J Health Syst Pharm. 2017 Sep 15;74(18):1405-1411. doi: 10.2146/ajhp170025. PMID 28887342
- [Background] Zarobe L, Bungay H. The role of arts activities in developing resilience and mental wellbeing in children and young people a rapid review of the literature. Perspect Public Health. 2017 Nov;137(6):337-347. doi: 10.1177/1757913917712283. Epub 2017 Jun 14. PMID 28613107
- [Background] Ali A, Wolfert S. Theatre as a treatment for posttraumatic stress in military veterans: Exploring the psychotherapeutic potential of mimetic induction. The Arts in Psychotherapy 50: 58-65, 2016.
- [Background] Bennington R, Backso A, Harrison J, Reader AE, Carolan R. Art therapy in art museums: Promoting social connectedness and psychological well-being of older adults. The Arts in Psychotherapy 49: 34-43, 2016.
- [Background] Coholic D, Eys, M, Lougheed S. Investigating the effectiveness of an arts-based and mindfulness-based group program for the improvement of resilience in children in need. Journal of Child & Family Studies 21(5): 833-844, 2011.
- [Background] Czamanski-Cohen J, Sarid O, Huss E, Ifergane A, Niego L, Cwikel J. CB-ART: The use of a hybrid cognitive behavioral and art based protocol for treating pain and symptoms accompanying coping with chronic illness. The Arts in Psychotherapy 41: 320-328, 2014.
- [Background] Ernestus SM, Prelow HM. Patterns of risk and resilience in African American and Latino Youth. Journal of Community Psychology 43(8): 954-972, 2015.
- [Background] An assessment of the value of music therapy for haemato-oncology patients. Cancer Nursing Practice 13(5): 22-28, 2014.
- [Background] Hill CA, Gunderson CJ. Resilience of lesbian, gay, and bisexual individuals in relation to social environment, personal characteristics, and emotion regulation strategies. Psychology of Sexual Orientation & Gender Diversity 2(3): 232-252, 2012.
- [Background] Kaimal G, Gonzaga AML, Schwachter V. Crafting, health, and wellbeing: Findings from the survey of public participation in the arts and considerations for art therapists. Arts & Health 9(1): 81-90, 2017.
- [Background] Kindig D, Stoddart G. What is population health? Am J Public Health. 2003 Mar;93(3):380-3. doi: 10.2105/ajph.93.3.380. PMID 12604476
- [Background] Letwin L, Silverman MJ. No between-group difference but tendencies for patient support: A pilot study of a resilience-focused music therapy protocol for adults on a medical oncology/hematology unit. The Arts in Psychotherapy 55: 116-125, 2017.
- [Background] Pasiali V. Resilience, music therapy, and human adaptation: Nurturing young children and families. Nordic Journal of Music Therapy 21(1): 36-56, 2012.
- [Background] Rankanen M. Clients' experiences of the impacts of an experiential art therapy group. The Arts in Psychotherapy 50: 101-110, 2016.
- [Background] Sabogal M. Community arts in the lives of disadvantaged African American youth: Educating for wellness cultural praxis. (Doctoral dissertation). Retrieved from ProQuest, LLC (3587830), 2013.
- [Background] Shim M, Johnson RB, Gasson S, Goodill S, Jermyn R, Bradt J. A model of dance/movement therapy for resilience-building in people living with chronic pain. European Journal of Integrative Medicine 9: 27-40, 2017.
- [Background] Sung H-K. The influence and role of arts on community well-being. (Unpublished doctoral dissertation). Arizona State University, Tempe, AZ, 2016.